CLINICAL TRIAL: NCT03393767
Title: Time Course of Activity Signs at High Resolution OCT During OCT-guided High Frequency Intravitreal Ranibizumab Treatment in Choroidal Neovascularization Due to Age Related Macular Degeneration
Brief Title: Time Course of Activity Signs at SD-OCT High Frequency Intravitreal Ranibizumab Treatment in CNV Due to AMD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vista Klinik (Other)
Responsible Party: Principal Investigator, Dr. med. Katja Hatz, Prof. Christian Pruente, Vista Klinik
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OCT-2010-07
Record Dates: First submitted 2014-11-26; First posted 2018-01-08 (Actual); Last update posted 2018-01-08 (Actual); Status verified 2018-01

CONDITIONS: Choroidal Neovascularization; Age Related Macular Degeneration
Keywords: CNV; AMD; ranibizumab
MeSH Terms: conditions — Choroidal Neovascularization; Macular Degeneration | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- prospective 1- Arm (Other): OCT-guided high frequency intravitreal ranibizumab 0.5mg
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab — Intravitreal injection
  Other Names: Lucentis

SUMMARY:
The purpose of the study is to detect persisting or early new activity of choroidal neovascularization (CNV) due to age related macular degeneration (AMD) during the first 12 months following the first ranibizumab dose at baseline as assessed by weekly high resolution optical coherence tomography (OCT). Detection of persisting or new signs of CNV activity at OCT triggers further ranibizumab treatments considering that any ranibizumab injections can maximally be applied as often as 2-weekly.

DETAILED DESCRIPTION:
This is a prospective, 1-arm, monocenter study designed to evaluate the time course of early re-activation of CNV assessed by High Resolution OCT. An OCT-guided high frequency (up to 2-weekly) intravitreal ranibizumab treatment in CNV due to AMD may prevent further growth and early re-growth of CNV as evaluated by OCT at a weekly basis.

Consenting, enrolled patients will receive one 0.5 mg ranibizumab intravitreal injection at baseline (month 0). Afterwards all patients will undergo a weekly OCT assessment. Further treatments, which can maximally be applied as often as 2-weekly, are triggered by persisting or new signs of CNV activity at OCT as defined by intraretinal cysts or subretinal fluid. For this study, a month is defined as 28 days, a 2-week period as 14 days. During the 12-month study period, a maximum of 24 ranibizumab injections may be administered.

An interim analysis will not be performed. The study will be conducted in compliance with the protocol, GCP and the applicable regulatory requirement(s).

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥ 50 years of age.
* Patients with active primary subfoveal CNV secondary to AMD, including those with predominantly classic, minimally classic or occult lesions with no classic component.
* Evidence that CNV extends under the geometric center of the foveal avascular zone.
* Total CNV area encompassed within the lesion must be ≥ 50% of total lesion area.
* The total lesion area ≤ 12 disc areas for minimally classic or occult with no classic component and ≤ 9 disc areas (5400µm) in greatest linear dimension with predominantly classic lesions.
* Patients who have a BCVA of 20/32 to 20/320 (letter score of 78 to 25 letters) in the study eye using ETDRS charts.
* Willing and able to give written informed consent according to legal requirements, and who have signed the consent form prior to initiation of any study procedure.
* Willing and able to comply with study procedures.

Exclusion Criteria:

* Subretinal hemorrhage in the study eye that involves the center of the fovea, if the size of the hemorrhage is either ≥ 50% of the total lesion area or ≥ 1 disc area in size.
* Structural damage to the center of the macula (beside CNV) in the study eye.
* Presence of a retinal pigment epithelial tear involving the macula in the study eye.
* Patients with angioid streaks or precursors of CNV in either eye due to other causes.
* Concurrent disease in the study eye that could compromise visual acuity or require medical or surgical intervention during the 12-month study period.
* Vitreous hemorrhage, history of rhegmatogenous retinal detachment or macular hole.
* Active intraocular inflammation (grade trace or above) in the study eye.
* Any active infection involving ocular adnexa.
* History of uncontrolled glaucoma in the study eye.
* Aphakia with absence of the posterior capsule in the study eye.
* Any prior treatment in the study eye with verteporfin, subfoveal focal laser photo-coagulation, vitrectomy, transpupillary thermotherapy, intravitreally applied drugs.
* History of submacular surgery or other surgical intervention for AMD in the study eye.
* Extracapsular extraction of cataract within 3 months preceding Baseline.
* Previous violation of posterior capsule in the study eye (unless YAG capsulotomy).
* History of Stroke.
* Pregnant or nursing (lactating) women.
* History of hypersensitivity or allergy to fluorescein.
* Inability to obtain OCT/photographs/fluorescein angiograms of sufficient quality.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-12; Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in CNV activity (any fluid) as assessed by High Resolution OCT | 12 month OCT Assessment
  The primary objective is to evaluate the time course of early re-activation of CNV assessed by High Resolution OCT.

SECONDARY OUTCOMES:
To evaluate the correlation between activation of CNV evaluated by OCT (any fluid) and changes of BCVA. | 12 month
  ► To evaluate the correlation between activation of CNV evaluated by OCT (any fluid) and changes of BCVA.
To evaluate the effect of OCT-guided up to 2-weekly dosing of ranibizumab on BCVA changes at month 12. | 12 months
  To evaluate the effect of OCT-guided up to 2-weekly dosing of ranibizumab on BCVA changes at month 12.
To evaluate the effect of OCT-guided up to 2-weekly dosing of ranibizumab on the total number of injections needed within the 12 months observation period. | 12 months
  To evaluate the effect of OCT-guided up to 2-weekly dosing of ranibizumab on the total number of injections needed within the 12 months observation period.
To evaluate the safety and tolerability of up to 2-weekly dosing of ranibizumab by determining the rates of adverse events and serious adverse events at month 12. | 12 months
  To evaluate the safety and tolerability of up to 2-weekly dosing of ranibizumab by determining the rates of adverse events and serious adverse events at month 12.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Pruente, MD, Principal Investigator — Vista Klinik
Locations (1):
- Vista Klinik, Binningen, Switzerland